CLINICAL TRIAL: NCT01084733
Title: Correlative Study of Nicotine Levels With Response Rates to Therapy Using Radiation Alone or in Combination With Chemotherapy in Head and Neck Cancer
Brief Title: Nicotine Levels With Response Rates to Radiation Alone or With Chemo In Head & Neck Cancer
Status: Completed | Type: Observational
Sponsor: Mahesh Kudrimoti (Other)
Responsible Party: Sponsor-Investigator, Mahesh Kudrimoti, Clinical Faculty, Radiation Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: MCC-06-0781-P3K; NICOTINE-HN (Other: Markey Cancer Center)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Larynx Cancer; Lip Cancer; Oral Cavity Cancer; Pharyngeal Cancer; Oropharyngeal Cancer
MeSH Terms: conditions — Laryngeal Neoplasms; Lip Neoplasms; Mouth Neoplasms; Pharyngeal Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be obtained weekly during the treatment phase. Serum will be collected and aliquoted into eppendorf tubes. Serum samples will be stored in -20C freezer until assayed for cotinine levels using Immulite immunoassay for cotinine (Immulite 2000 Assay, DPC, United States, Technical Services 800-372-1782).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to evaluate the relationship between serum nicotine levels and tumor response of squamous cell cancers of the head and neck (SCCHN) to radiotherapy alone or in combination with chemotherapy.

Correlation of RECIST response, volumatic response, pathologic response (in patients receiving post-treatment neck dissection), and hemodynamic response (tumor oxygenation and blood flow) will be performed.

DETAILED DESCRIPTION:
The exposure to tobacco related carcinogens is highly dependent upon dose as well as interindividual characteristics of metabolism. Risk assessment of carcinogenic profiles for nicotine and its individual metabolites is complicated by interindividual variations in nicotine metabolism associated with quantitative nicotine exposure, gender, genetic polymorphisms, and behavioral and environmentally induced differences in nicotine metabolizing enzyme activities. Consequently, differences in smoking behavior or tobacco use have been correlated to differences in nicotine metabolism resulting in cessation strategies based upon tobacco use, nicotine dependence, and behavioral modification. Cotinine has been shown to be a reliable marker of nicotine exposure and more reflective of recent rather than acute nicotine use with better assessment of baseline nicotine levels. Therefore, subjects will have blood samples drawn weekly during radiation for cotinine analysis.

Radiation therapy efficacy is known to be dependent on tissue oxygen status. Since therapeutic treatment is less efficacious in patients with poorly vascularized/ hypoxic tumors, it is desirable to identify and target such patients for special treatment. Recent magnetic resonance imaging and computed tomography investigations have shown that there are significant blood flow changes during radiation or chemo-radiation therapy, suggesting that early blood flow may have prognostic value. Among those methods for oxygen and blood flow measurements, the near-infrared spectroscopy (NIRS) is more benefit with merit of non-invasive, portable, fast test, and inexpensive. Our instrument system combined near-infrared diffuse reflectance spectroscopy (DRS) and diffuse correlation spectroscopy (DCS) is capable of monitoring tissue oxygen and blood flow simultaneously. This hybrid diffuse optical instrument has already been used for monitoring of therapeutic effects (e.g., radiation therapy, chemotherapy) in tumors in human head & neck and breast. In this study, we will use this hybrid instrument to investigate the hemodynamic responses to different therapies (radiation alone, radiation + chemotherapy) in patients with different nicotine levels. Baseline measurement of tissue oxygen saturation, total hemoglobin concentration and blood flow using a hybrid optical instrument (DRS for oxygen measurement and DCS for blood flow measurement). A hand-hold optical probe connected to the hybrid instrument will be placed on the head/neck tumor for about 3-5 minutes, then move it on the normal arm muscle for control purposeTumor oxygenation and flow measurements will be performed at the beginning of every week during the treatment period. During this monitoring process non-invasive blood pressure monitoring will also occur. Weekly optical measurements will be obtained during treatment.In this study we will investigate the hemodynamic responses to different nicotine levels and different therapies (radiation alone, radiation + chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* A: Male or female aged 18 or older
* B: Pathologically confirmed squamous cell carcinoma
* C: Measurable disease using CT, MRI, or panendoscopy
* D: Tumor sites to include:

Oropharynx Hypopharynx Oral cavity Larynx Measurable disease with no evidence of primary

* E: Patients to be treated with radiotherapy or chemoradiotherapy as a primary treatment modality. Patients to be treated with radiotherapy in combination with platinum based chemotherapy will be considered for enrollment.
* F: Nutritional status to include patients that do not require placement of a feeding tube as well as patients that are feeding tube dependent. However, patients requiring total parenteral nutrition prior to initiation of treatment will be excluded.
* G: ECOG performance status of 0, 1 or 2.
* H: Standard of care chemotherapy inclusion criteria to include:

  i: No evidence of active angina pectoris or ventricular arrhythmia's; no myocardial infarction within the last six months. (Patients with medically controlled hypertension or congestive heart failure are eligible.) ii: Absolute neutrophil count of > 1000/uL and platelet count > 100,000/uL iii: Serum total bilirubin < 1.5 mg/dL iv: Creatinine Clearance greater than 60 ml/min creatinine clearance to be calculated using the formula: (140 - age) x (wgt in kg) * (serum creatinine) x (72)

  * multiply by 0.85 for females v: If a pre-existing grade I neuropathy exists, patients must be willing to risk worsening neuropathy secondary to treatment. Patients with grade II or greater neuropathy will be excluded from study.
* I: Standard of care treatment will require counseling against the use of tobacco products and can include nicotine replacement at the request of the patient and discretion of treating physician. Patients who continue to use tobacco products as well as patients using any form of cessation strategy (nicotine replacement, bupropion, or other) will be eligible for enrollment.
* J: Patients enrolled on experimental studies will be considered for enrollment with final selection to be made by Dr. Kudrimoti, Dr. Warren, Dr. Arnold, and Dr. Valentino.
* K: Ability to give informed consent

Exclusion Criteria:

* A: Pregnant females. Males and females of childbearing potential must use effective contraception in order to prevent pregnancy during therapy.
* B: Histology other than squamous cell carcinoma
* C: Patients without measurable disease using CT, MRI, or panendoscopy
* D: Patients eligible for surgical resection alone or with significant (> 25%) surgical tumor debulking prior to radiotherapy will not be considered for enrollment. Furthermore, patients who are otherwise not candidates for radiotherapy at the discretion of the treating physician will be excluded from enrollment.
* E: Patients with a history of previous or current malignancy at other sites diagnosed within the last 5 years, with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain free of recurrence or metastases for greater than five years are eligible.
* F: Patients with active infection will not be eligible for this protocol until the infection is treated and the symptoms have clinically resolved.
* G: Prior chemotherapy, prior irradiation or surgery for SCCHN will not be allowed.
* H: Patients with metastatic disease will not be eligible for this study.
* I: Patients with grade II or greater peripheral neuropathy will be excluded from study.
* J: Patients receiving medication to prevent mucositis (palifermin, amifostine, or other).
* K: Patients requiring total parenteral nutritional support prior to the initiation of treatment will not be eligible for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female aged 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2007-08; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation of serum cotinine with volumetric response | 2 years from start of treatment
  RECIST criteria will be used as a correlate for standardization of tumor response. Volumetric analysis may provide better assessment of bulky tumor size that may have a large necrotic or hypoxic component that may be resistant to treatment. Furthermore, volumetric analysis has been associated with a higher rate of concordance to response based upon RECIST criteria.

SECONDARY OUTCOMES:
Correlation of serum cotinine with toxicities during treatment. | 90 days from start of treatment
  Toxicities will be graded using the National Cancer Institute (NCI) scale for acute and subacute toxicity and the Radiation Therapy Oncology Group's late toxicity scale.
Correlation of serum cotinine with time to progression. | 2 years
  Time to progression will be calculated as the time interval between the start of radiation treatment and the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Correlation of serum cotinine with survival | 5 years from start of treatment
  Survival will be calculated from the start of radiation to the date of death.
Correlation of serum cotinine with response to treatment | 5 years
  Both pathologic and radiographic response to therapy will be assessed where possible. Primary tumors will be assessed by the attending otolaryngologist by panendoscopy, with biopsies taken in the case of a question of response. Nodal disease response will be assessed by radiographic means. All patients will be assessed for response at the end of primary treatment.
Investigate the hemodynamic responses to different nicotine levels and different therapies (radiation alone, radiation + chemotherapy). | End of Treatment
  Previous studies indicated that there is a significant increase in blood flow in the early two weeks of radiation therapy and decreases in the following weeks, while the tissue oxygen saturation tends to decline continually

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Kudrimoti, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No